CLINICAL TRIAL: NCT04176835
Title: Neurobiological Effects of Oxytocin on Social Decision Making in Schizophrenia: A Pharmacological MRI Study
Brief Title: Oxytocin and Social Decision Making in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dr Naren P Rao, Additional Professor of Psychiatry, National Institute of Mental Health and Neuro Sciences, India
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 00861
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin (Experimental): Single-dose intranasal oxytocin or intranasal placebo administered in counterbalanced order
  Interventions: Drug: Oxytocin nasal spray
- Placebo (Placebo Comparator): Single-dose intranasal oxytocin or intranasal placebo administered in counterbalanced order
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — Single-dose oxytocin will be administered intranasally
  Arms: oxytocin
Drug: Placebo
  Arms: Placebo

SUMMARY:
schizophrenia patients and healthy volunteers will be included. Subjects who meet the inclusion and exclusion criteria for the study will be recruited. After completion of clinical assessments and neuropsychological assessments, all subjects will undergo two fMRI scans. In one scan subjects will receive a single dose of intranasal oxytocin and in another scan, they will receive intranasal saline. The order of administration of oxytocin or saline will be counterbalanced so that they are not administered in the same order to all subjects. Subjects will be blind to the drug administered.

ELIGIBILITY:
Schizophrenia group -

Inclusion Criteria:

1. Males between 18 and 45 years with at least 7 years of education
2. The DSM-IV diagnosis of Schizophrenia or schizoaffective or schizophreniform disorder
3. capacity to provide informed consent

Exclusion Criteria:

1. Current comorbid DSM-IV axis I diagnosis
2. General impaired intellectual functioning
3. history of alcohol or substance abuse or dependence in the last 12 months
4. contraindication to Oxytocin like hypersensitivity, vascular disease, chronic nephritis, epilepsy, asthma
5. past history of head injury resulting in loss of consciousness or neurosurgery
6. concomitant severe medical conditions
7. metal implants or paramagnetic objects within the body or claustrophobia which may interfere with the MRI.

Healthy volunteers:

Inclusion Criteria:

1. Males between 18 and 45 years with at-least 7 years education
2. Capacity to provide informed consent
3. absence of past or present psychiatric illnesses including substance abuse/dependence

Exclusion criteria:

1. General impaired intellectual functioning
2. contraindication to Oxytocin like hypersensitivity, vascular disease, chronic nephritis, epilepsy, asthma
3. past history of head injury resulting in loss of consciousness or neurosurgery
4. concomitant severe medical conditions
5. metal implants or paramagnetic objects within the body or claustrophobia which may interfere with the MRI.
6. Family history of schizophrenia or schizoaffective or schizophreniform disorder in a first-degree relative

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
fMRI changes with oxytocin while performing ultimatum game and at rest | 90 minutes
  Changes in brain activity and functional connectivity

IPD SHARING:
Plan to Share IPD: No